CLINICAL TRIAL: NCT02342600
Title: SARC029: Phase II Pilot Study of Trametinib in Combination With Pazopanib in Patients With Metastatic or Local-regionally Recurrent GIST (Gastrointestinal Stromal Tumor) Refractory or Intolerant to at Least Imatinib and Sunitinib
Brief Title: SARC029: Trametinib and Pazopanib in Patients With GIST (Gastrointestinal Stromal Tumor)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Supporting company withdrew interest
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC029
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-03

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — pazopanib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trametinib with Pazopanib (Experimental): Participants will take pazopanib (800mg) and trametinib (2mg) by mouth daily for a 28 day cycle.
  Interventions: Drug: Pazopanib; Drug: Trametinib

INTERVENTIONS:
Drug: Pazopanib — A kinase inhibitor indicated for the treatment of patients with advanced renal cell carcinoma and advanced soft tissue sarcoma who have receive prior chemotherapy.
  Other Names: Votrient
Drug: Trametinib — A kinase inhibitor indicated for the treatment of patients with unresectable or metastatic melanoma with BRAF V600E or V600K mutations as detected by an FDA-approved test.
  Other Names: Mekinist

SUMMARY:
This study evaluates the combination of trametinib and pazopanib in patients with advanced gastrointestinal stromal tumors (GIST).

DETAILED DESCRIPTION:
Trametinib and pazopanib are independently approved for other cancers. Both drugs work to inhibit tumor development in different ways. Combining these drugs may lead to improved disease control. The purpose of this study is to evaluate the effect of the combination of both drugs on advanced gastrointestinal stromal tumors.

ELIGIBILITY:
Inclusion Criteria includes:

* Age ≥ 18 years
* Histologically confirmed diagnosis of advanced GIST
* ECOG performance status of 0-1
* Measurable disease as per modified RECIST 1.1
* Prior disease progression on at least imatinib and sunitinib. Maximum of 3 prior kinase inhibitors allowed for treatment of advanced disease. Patients with prior exposure to pazopanib or MEK inhibitors are not eligible.
* Adequate organ systems function within 14 days (and 72 hours) prior to start of protocol therapy
* Patients must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up.
* Women of childbearing potential must have a negative urine or blood pregnancy test within 7 days of Cycle 1 Day 1. Fertile men and women of childbearing potential must agree to use effective contraception as defined in Section 7 during the study and for 4 months following the last dose of study drugs in both sexes.
* Life expectancy of ≥ 3months

Exclusion Criteria includes:

* Prior malignancy.
* Central nervous system (CNS) metastases at baseline, with the exception of those patients who have previously-treated CNS metastases (surgery +/- radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria:

are asymptomatic and have no requirement for steroids or enzyme-inducing anticonvulsants in at least 3 months prior to screening.

* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
* QTcB interval > 480 msec
* History of one or more of the following cardiovascular conditions within the past 6 months:

Cardiac angioplasty or stenting Myocardial infarction Unstable angina Coronary artery bypass graft surgery Symptomatic peripheral vascular disease Class II, III, or IV congestive heart failure, as defined by the New York Heart Association (NYHA) Uncontrolled arrhythmias

* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥ 140 mm Hg or diastolic blood pressure (DBP) of ≥ 90 mmHg].
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement are not considered to be major surgery).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.
* Recent hemoptysis (≥ 1/2 teaspoon of red blood within 8 weeks before first dose of study drug)
* Any serious and or unstable pre-existing medical, psychiatric, or other condition that could interfere with the patient's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications listed in Section 5.2.4 for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Treatment with any of the following anti-cancer therapies:
* Radiation therapy or tumor embolization within 14 days prior to the first dose of OR
* Chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug.
* Ipilimumab must have been discontinued at least 8 weeks prior to initiation of treatment with trametinib
* Administration of any non-oncologic investigational drug within 30 days or five half-lives (whichever is longer) prior to the first dose of study drug.
* Any ongoing toxicity from prior anti-cancer therapy that is ≥ Grade 1 and/or that is progressing in severity, except alopecia.
* Inability to swallow and retain oral medication
* Known or suspected allergy or hypersensitivity to pazopanib, trametinib (GSK1120212), or excipients of the formulations given during the course of this trial.
* History of interstitial lung disease or pneumonitis, intracardiac defibrillators, known HIV, active HBV or HCV infections, history of retinal vein occlusion, symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 16 weeks
  Disease Control Rate (DCR) is the percentage of patients who have achieved complete response, partial response and stable disease to study treatment

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 12 months
  Date of first dose of drug to date of imaging demonstrating disease progression.
Overall Survival (OS) | up to 10 years
  Time from first date of drug administration to date of death from any cause
Number and type of adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Ganjoo, MD, Principal Investigator — Stanford University

REFERENCES:
- See also: Sarcoma Alliance for Research through Collaboration — http://www.sarctrials.org/sarc-clinical-trials